CLINICAL TRIAL: NCT03785769
Title: Effect of Pre-etching of Dentin on Survival of Restorations With High Viscosity Glass Ionomer Cement in the Atraumatic Restorative Treatment - Randomized Clinical Trial Restorations With High Viscosity Glass Ionomer Cement
Brief Title: Pre-etching of Dentin Before Restorations With High Viscosity Glass Ionomer Cement
Acronym: CEPECO4
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Outbreak of COVID-19.
Sponsor: Universidade Ibirapuera (Other)
Responsible Party: Principal Investigator, Tamara Kerber Tedesco, Principal investigator, Universidade Ibirapuera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Unib4
Record Dates: First submitted 2018-12-18; First posted 2018-12-24 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind (Patient and Examiner) will not be able to blinding the operator due to the obvious difference between the techniques
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVGIC restoration with pre-etching (Active Comparator): Pre-etching of the surface with polyacrylic acid for 10 s, followed by HVGIC restoration.
  Interventions: Procedure: HVGIC restoration with pre-etching
- HVGIC restoration with non pre-etching (Experimental): HVGIC restoration without the pre-etching of the surface.
  Interventions: Procedure: HVGIC restoration with non pre-etching

INTERVENTIONS:
Procedure: HVGIC restoration with pre-etching — Pre-etching of the surface with polyacrylic acid for 10 s, followed by washing and drying the cavity with cotton balls; and fill with HVGIC, inserted into the cavity with the aid of an insertion spatula and adapted to the cavity by the digital pressure technique.
  Arms: HVGIC restoration with pre-etching
Procedure: HVGIC restoration with non pre-etching — Restoration with HVGIC, inserted into the cavity with the aid of an insertion spatula and adapted to the cavity by the digital pressure technique.
  Arms: HVGIC restoration with non pre-etching

SUMMARY:
The objective of this randomized clinical trial is to evaluate the survival of restoration with high viscosity glass ionomer cement (HVGIC) with pre-etching with polyacrilic acid compared with no pre-etching in order to treat occlusoproximais caries lesion in primary molars, as well as the impact of those treatments in the caries lesion progression, the cost-efficacy of the procedures and the discomfort reported by the patient. Children of 4 to 8 years will be selected in the Pediatric Dentistry Clinic of Universidade Ibirapuera. 192 teeth will be randomized in 2 experimental groups: (1) HVGIC restoration with pre-etching and (2) HVGIC restoration with no pre-etching. Will be considered as primary outcome the survival of the restoration evaluated after 6, 12, and 24 months by two trained examiners. The carious lesions progression will be evaluated after 24 months of follow-up. The time of the treatments and the cost of the materials will be considered to estimate the cost-efficacy of each treatment. The discomfort reported by the participant will be measured after each procedure following the Wong-Baker scale. For the primary outcome, Kaplan-Meier survival and the Long-Rank test will be used in order to compare the two groups. Cox regression will be performed in order to evaluate thee influence of explanatory variables on the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carious lesion of occlusoproximais in primary molars

Exclusion Criteria:

* Patients will be excluded with special needs, using orthodontics devices and/or systemic diseases which may affect the oral cavity.
* Also, teeth with pulp exposure, spontaneous pain, mobility, presence of abscess or fistula next to the tooth, teeth with restorations, sealants or enamel formation defects will also be excluded.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival of restorations | 24 months
  Comparing the survival of HVGIC restorations without pre-etching with HVGIC restorations with pre-etching by clinical assessment using a criteria proposed by Roleveld et al., 2006.

SECONDARY OUTCOMES:
Caries lesion progression will be evaluated by comaparison of radiograph immediately after the restoration | Immediately after the restoration and 24 months
  The caries lesion progression will be evaluated by comaparison of radiograph immediately after the restoration and after 24 months.
Cost-efficacy | 24 months.
  The duration of the treatments (time of treatment) and the cost of the materials used will be considered for the estimation of the cost-efficacy of the treatments by a ratio - cost/efficacy, being efficacy considered the tooth survival.
Discomfort regarding the treatment options by a Wong-Baker FACES pain rating scale | Immediately after the treatment
  Children-reported discomfort regarding the treatment options by a Wong-Baker FACES pain rating scale. The scale present 6 different faces since "very happy" until "very sad" with the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tamara Kerber Tedesco, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available on Mendeley database.